CLINICAL TRIAL: NCT03985956
Title: The Validity and Reliability of the ADL-Glittre Test as a Measure of Functional Capacity in Children With Asthma
Brief Title: Pediatric Glittre ADL-test in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, PhD, PT, Research Assistant, Gazi University
Other Study IDs: 13579
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Asthma in Children
Keywords: Daily Living Activities; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate reliability, validity, of the Glittre ADL Test in children with Asthma.

DETAILED DESCRIPTION:
The TGlittre-P is an adaptation of the TGlittre test for pediatric patients. It consists of completing a circuit while carrying a backpack with a variable weight of 0.5 kg to 2.5 kg, according to the child´s age and sex. This weight range follows the guidelines of the World Health Organization, which states that the younger the female child is, the lighter the backpack should be, in order to assure the school children´s health condition. The following tasks should be carried out; from a sitting position, the child stands up and walks along a 10m-long flat course, going up and down a 2-step rise (17 cm high x 27 cm wide) about halfway along that distance, to reach a bookshelf with three 0.5 kg objects (i.e. colorful plastic bowling pins filled with sand). The objects are placed on the top shelf at eye level, which should be removed, one by one, to the lower shelf at the level of the umbilicus, and then to the ground. Next, the objects should be placed on the lower shelf and then back to the top shelf. The child walks back along the same route. (S)he sits down, stands up and immediately starts the next lap. The following verbal instructions are given during the test: "sit" and "stand." The time required to walk five laps is registered; the less the time spent, the better the performance is. The test performance was evaluated by comparing the patient´s data with the data predicted by the equation, in his study with healthy children. The equation for girls is "time in TGlittre-P = 3.781-0.083 x AGE"; and boys, "time in TGlittre-P = 4.025-0.123 x AGE".

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6-14 years with a diagnosis of Asthma
* Task-oriented and co-operative patients without any musculoskeletal, rheumatic, neurological, hearing and visual diseases and without pulmonary exacerbation at the time of data collection will be included in this study.

Exclusion Criteria:

-

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with asthma who apply to Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Glittre ADL test | 15 minutes
  Functional test

SECONDARY OUTCOMES:
Six Minute Walk Test | 10 mimutes
  Exercise Test

CONTACTS AND LOCATIONS:
Overall Officials: Müşerrefe N Keleş, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)